CLINICAL TRIAL: NCT02578238
Title: Post-Marketing Surveillance of Humira in Korean Pediatric CD Patients Under the "New-Drug Re-examination"
Brief Title: Post-Marketing Surveillance of Humira in Korean Pediatric Crohn's Disease (CD) Patients Under the "New-Drug Re-examination"
Status: Completed | Type: Observational
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Other Study IDs: P15-619
Record Dates: First submitted 2015-10-15; First posted 2015-10-16 (Estimated); Results first posted 2018-12-19 (Actual); Last update posted 2018-12-19 (Actual); Status verified 2018-05

CONDITIONS: Pediatric Crohn's Disease
Keywords: Korea; Humira; Pediatric Crohn's Disease
MeSH Terms: conditions — Pediatric Crohn's disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Participants With Pediatric CD: Participants with pediatric CD who have been prescribed Humira® (adalimumab) by the treating physician.

SUMMARY:
This study is a non-interventional, observational study of Humira® in the treatment of pediatric CD as per the New Drug Re-examination Guideline in Korea. This study will be conducted in institutions which provide a written agreement to AbbVie Korea, and where the use of Humira® for pediatric CD is following their normal medical practice setting. Pediatric patients who are prescribed Humira® as per physician's medical judgment in accordance with the approved Korean local label will be enrolled in the study. As this is a post marketing surveillance, AbbVie is NOT involved in the product supply since the drug is being used according to the approved marketing label and is to be prescribed by the physician under usual and customary practice of physician prescription.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric patients with CD who are prescribed Humira in accordance with the Korean label for Humira authorization (labeling)
* Patients who have given written authorization to use their personal health data for the purposes of this study.

Exclusion Criteria:

* Any contraindications to Humira as listed on the approved product market authorization (labeling)
* Patients who is participating on other clinical trials.

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Pediatric CD patients who have been prescribed Humira® by the treating physician
Sampling Method: Probability Sample
Enrollment: 143 (Actual)
Dates: Start 2015-09-24 (Actual); Primary Completion 2017-05-31 (Actual); Study Completion 2017-05-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eunjung Gu, MS, Study Director — AbbVie korea

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Regarding Medicine Information — http://rxabbvie.com/

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Case report forms were retrieved from 152 participants during the study period. Among these participants, 143 were included in the safety analysis population, excluding 9 participants who did not use the drug according to the approved indication or dosage.
Groups:
- Participants With Pediatric Crohn's Disease (CD): Participants with pediatric CD prescribed Humira® by their treating physician.
Period: Overall Study
Arm/Group | Participants With Pediatric Crohn's Disease (CD)
Started | 143
Completed | 143
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Participants With Pediatric Crohn's Disease (CD)
Number analyzed (Participants) | 143
Age, Continuous [Mean (Standard Deviation); unit: years] | 14.14 (2.43)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 56
  Male | 87
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Korean | 143

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Adverse Events (AEs)/Adverse Drug Reactions (ADRs), Serious AEs/ADRs and Unexpected AEs/ADRs
Description: An AE is defined as any untoward medical occurrence, which does not necessarily have a causal relationship with their treatment. If an AE meets any of the following criteria, it is considered a serious AE: results in death, is life-threatening, results in hospitalization or prolongation of hospitalization, is a congenital anomaly, results in persistent or significant disability/incapacity, is an important medical event requiring medical or surgical intervention to prevent serious outcome. An ADR label was used for an AE when causal relationship with a pharmaceutical drug could not be excluded.
Time Frame: From Day 0 (informed consent) to up to 70 days following the last administration of Humira®. The mean length of treatment was 52.81 (±45.58) weeks (calculated based on participants with available start date data [n=142]).
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Participants With Pediatric Crohn's Disease (CD)
Number analyzed (Participants) | 143
percentage of participants
  AEs | 18.18 [12.23 to 25.49]
  ADRs | 14.69 [9.33 to 21.57]
  Serious AEs | 5.59 [2.45 to 10.73]
  Serious ADRs | 3.50 [1.14 to 7.97]
  Unexpected AEs | 6.29 [2.92 to 11.61]
  Unexpected ADRs | 2.80 [0.77 to 7.01]

ADVERSE EVENTS:
Time Frame: From Day 0 (informed consent) to up to 70 days following the last administration of Humira®. The mean length of treatment was 52.81 (±45.58) weeks (calculated based on participants with available start date data [n=142]).
Groups:
- Participants With Pediatric CD: Participants with pediatric CD prescribed Humira® by their treating physician.
Arm/Group | Participants With Pediatric CD
All-Cause Mortality (participants affected / at risk) | 0/143
Serious Adverse Events (participants affected / at risk) | 8/143
Other Adverse Events (participants affected / at risk) | 22/143
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Participants With Pediatric CD (N=143)
Abdominal pain (Gastrointestinal disorders) | 2
Gastrointestinal necrosis (Gastrointestinal disorders) | 1
Haematochezia (Gastrointestinal disorders) | 1
Ileus paralytic (Gastrointestinal disorders) | 1
Intestinal obstruction (Gastrointestinal disorders) | 1
Intestinal perforation (Gastrointestinal disorders) | 1
Small intestinal obstruction (Gastrointestinal disorders) | 1
Appendicitis (Infections and infestations) | 1
Peritonitis (Infections and infestations) | 1
Pyrexia (General disorders) | 1
Candida infection (Infections and infestations) | 1
Pyelonephritis acute (Infections and infestations) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Participants With Pediatric CD (N=143)
Diarrhoea (Gastrointestinal disorders) | 2
Haematochezia (Gastrointestinal disorders) | 1
Intestinal stenosis (Gastrointestinal disorders) | 2
Colonic haematoma (Gastrointestinal disorders) | 1
Gastrointestinal inflammation (Gastrointestinal disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 3
Pruritus (Skin and subcutaneous tissue disorders) | 1
Skin reaction (Skin and subcutaneous tissue disorders) | 1
Urticaria (Skin and subcutaneous tissue disorders) | 1
Alanine aminotransferase increased (Investigations) | 3
Aspartate aminotransferase increased (Investigations) | 3
Liver function test abnormal (Investigations) | 1
Leukopenia (Blood and lymphatic system disorders) | 4
Helicobacter gastritis (Infections and infestations) | 1
Malaise (General disorders) | 1
Pain (General disorders) | 1
C-reactive protein increased (Investigations) | 1
Red blood cell sedimentation rate increased (Investigations) | 1
Injection site erythema (General disorders) | 1
Folliculitis (Infections and infestations) | 1
Anastomotic complication (Injury, poisoning and procedural complications) | 1
Dizziness (Nervous system disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-04-29): https://cdn.clinicaltrials.gov/large-docs/38/NCT02578238/Prot_SAP_000.pdf